CLINICAL TRIAL: NCT00000994
Title: A Placebo-Controlled Trial To Evaluate Azidothymidine (AZT) in the Treatment of Human Immunodeficiency Virus (HIV) Infection in Patients With AIDS-Associated Kaposi's Sarcoma
Brief Title: A Study of AZT in HIV-Infected Patients With AIDS-Related Kaposi's Sarcoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: Double | Purpose: Treatment
Other Study IDs: ACTG 001; 10977 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: AIDS-Related Opportunistic Infections; Sarcoma, Kaposi; Acquired Immunodeficiency Syndrome; Zidovudine
MeSH Terms: conditions — HIV Infections; AIDS-Related Opportunistic Infections; Sarcoma, Kaposi; Acquired Immunodeficiency Syndrome | interventions — Zidovudine

INTERVENTIONS:
Drug: Zidovudine

SUMMARY:
To determine whether taking zidovudine (AZT) will change the natural course of HIV infection in patients with AIDS-associated Kaposi's sarcoma (KS) and whether administering AZT at a similar dose but at different intervals will reduce toxicity in a more manageable treatment plan.

Patients infected with AIDS can benefit from therapy with an effective anti-AIDS virus agent. AZT is a drug that is effective in inhibiting the effects of HIV infection. The study will show whether toxicity of AZT can be reduced in a more manageable treatment plan, and whether AZT therapy will delay the development of opportunistic infections and/or KS lesions.

DETAILED DESCRIPTION:
Patients infected with AIDS can benefit from therapy with an effective anti-AIDS virus agent. AZT is a drug that is effective in inhibiting the effects of HIV infection. The study will show whether toxicity of AZT can be reduced in a more manageable treatment plan, and whether AZT therapy will delay the development of opportunistic infections and/or KS lesions.

Patients are divided into two treatment groups, the first receiving AZT for 5 doses a day, and the second receiving AZT for 3 doses per day. A placebo group is divided into two to match the two treatment groups. Study patients are stratified according to whether they have (a) 10 or fewer cutaneous lesions without oral lesions or (b) more extensive cutaneous lesions or oral lesions. Patients are seen on an outpatient basis weekly for the first 2 months, every other week for the next 2 months, and monthly thereafter.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Acute treatment for mucocutaneous candidiasis, localized cutaneous herpes simplex, or localized or disseminated zoster infections.

Concurrent Treatment:

Allowed:

* Blood transfusion for treatment of Grade 3 hemoglobin toxicity if the patient's cardiovascular status is compromised or if the hemoglobin fails to show signs of recovery following withdrawal from the study drug. Toxicity grades according to NIAID Recommendations for Grading Acute and Subacute Toxic Effects (Adults).

Patients must have:

* HIV-related, biopsy-proven Kaposi's sarcoma mucocutaneous lesions without constitutional symptoms.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions will be excluded:

* Symptomatic, visceral Kaposi's sarcoma.
* Lymphedema.
* HIV neurologic disease as determined by a standard neurologic examination and neuropsychological questionnaire.

Concurrent Medication:

Excluded:

* Aspirin or acetaminophen on a regular basis or for longer than 72 hours without approval of investigator.
* Cimetidine.
* Flurazepam.
* Indomethacin.
* Ranitidine.
* Probenecid.
* Drugs causing anemia, neutropenia, or significant risk of nephrotoxicity.
* Prophylaxis or chronic suppression of herpes simplex.
* Treatment of herpes simplex virus cutaneous disease more often than once a month for 5 - 7 days.

Concurrent Treatment:

Excluded:

* Radiation therapy for treatment of Kaposi's sarcoma lesions.

The following patients will be excluded from the study:

* Patients with a history of any AIDS-defining opportunistic infection.
* Patients with any of the following constitutional symptoms with no etiology established:
* Temperature more than 38 degrees and/or drenching night sweats for more than 1 month; watery diarrhea for 2 or more weeks; weight loss of more than 10 percent.
* Patients with a history of other systemic malignancies or lymphomas.

Prior Medication:

Excluded:

* Systemic antineoplastic chemotherapy.
* Zidovudine (AZT).
* Excluded within 30 days of study entry:
* Antiretroviral agents.
* Immunomodulating agents.
* Prophylaxis for Pneumocystis carinii pneumonia.
* Prophylaxis for herpes simplex virus infections.
* Any other experimental therapy.

Prior Treatment:

Excluded within 30 days of study entry:

* Any experimental therapy.
* Active substance abuse.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240
Dates: Study Completion 1990-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Valentine FT, Study Chair
Locations (22):
- United States (22):
  - Los Angeles County - USC Med Ctr, Los Angeles, California
  - UCLA CARE Ctr, Los Angeles, California
  - Univ of California / San Diego Treatment Ctr, San Diego, California
  - San Francisco AIDS Clinic / San Francisco Gen Hosp, San Francisco, California
  - Stanford at Kaiser / Kaiser Permanente Med Ctr, San Francisco, California
  - Stanford Univ School of Medicine, Stanford, California
  - Charity Hosp / Tulane Univ Med School, New Orleans, Louisiana
  - Louisiana State Univ Med Ctr / Tulane Med School, New Orleans, Louisiana
  - Tulane Univ School of Medicine, New Orleans, Louisiana
  - Johns Hopkins Hosp, Baltimore, Maryland
  - Harvard (Massachusetts Gen Hosp), Boston, Massachusetts
  - Univ of Minnesota, Minneapolis, Minnesota
  - SUNY / Erie County Med Ctr at Buffalo, Buffalo, New York
  - City Hosp Ctr at Elmhurst / Mount Sinai Hosp, Elmhurst, New York
  - Beth Israel Med Ctr / Peter Krueger Clinic, New York, New York
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Mem Sloan - Kettering Cancer Ctr, New York, New York
  - Mount Sinai Med Ctr, New York, New York
  - Univ of Rochester Medical Center, Rochester, New York
  - SUNY / State Univ of New York, Syracuse, New York
  - Bronx Veterans Administration / Mount Sinai Hosp, The Bronx, New York
  - Duke Univ Med Ctr, Durham, North Carolina

REFERENCES:
- [Background] Chaisson RE, Fuchs E, Stanton DL, Quinn TC, Hendricksen C, Bartlett JG, Farzadegan H. Racial heterogeneity of HIV antigenemia in people with HIV infection. AIDS. 1991 Feb;5(2):177-80. doi: 10.1097/00002030-199102000-00007. PMID 1903261